CLINICAL TRIAL: NCT00321828
Title: A Phase II Trial of 5-Fluorouracil, Leucovorin, and Oxaliplatin (mFOLFOX6) Chemotherapy Plus Bevacizumab for Patients With Unresectable Stage IV Colon Cancer and a Synchronous Asymptomatic Primary Tumor
Brief Title: Combination Chemotherapy and Bevacizumab in Treating Patients With Stage IV Colon Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP C-10; U10CA012027 (NIH); CDR0000463513 (Other: NCI)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2013-01-14 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab (Experimental): Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — bevacizumab 5 mg/kg IV on day 1 every 14 days until excessive toxicity or disease progression
Drug: fluorouracil — 5-FU 400 mg/m2 IV bolus over 2-4 minutes then 2400 mg/m2 IV continuous infusion over 46 hours on day 1 every 14 days until excessive toxicity or disease progression
  Other Names: 5-FU
Drug: leucovorin — leucovorin 400 mg/m2 IV on day 1 every 14 days until excessive toxicity or disease progression
  Other Names: leucovorin calcium
Drug: oxaliplatin — Oxaliplatin 85 mg/m2 IV on day 1 every 14 days until excessive toxicity or disease progression

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colon cancer by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with bevacizumab works in treating patients with stage IV colon cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of major morbidity in patients with unresectable stage IV colon cancer and a synchronous asymptomatic primary tumor treated with fluorouracil, leucovorin calcium, and oxaliplatin (mFOLFOX6) in combination with bevacizumab without resection of the primary tumor.

Secondary

* Determine the rate of specific events related to the intact primary tumor requiring hospitalization or a major intervention but not requiring surgery.
* Determine the rate of ≥ grade 3 toxicity as defined by the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) that is related to study therapy prior to disease progression.
* Determine overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes, oxaliplatin IV given concurrently with leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years after study entry.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon

  * No histological findings other than adenocarcinoma of the colon
  * If the primary colon tumor and the metastatic lesions have been identified at the same time and it is not possible to biopsy the colonic lesion, the patient will be eligible without histologic confirmation of the primary cancer of the colon as long as other radiographic studies or scans document the characteristics of a colon cancer AND the biopsy of a metastatic site confirms diagnosis of adenocarcinoma suggestive of a primary tumor of the colon
* Unresected primary tumor of the colon AND radiographically confirmed metastatic colon cancer (single or multiple sites of metastases) that are not considered surgically resectable for cure by chest imaging and CT scan or MRI of the abdomen within the past 4 weeks and by endoscopy within the past 8 weeks
* Asymptomatic primary tumor

  * No obstruction, perforation, or active bleeding requiring transfusion
* Distal extent of the tumor must be ≥ 12 cm from the anal verge on endoscopy
* Not a candidate for curative surgical resection of all metastatic and colon primary tumors
* No evidence of Central Nervous System (CNS) metastases
* No recurrent local or metastatic disease after prior adjuvant therapy
* No diagnosis of rectal carcinoma

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count ≥ 1200/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN) (≤ 5.0 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 3.0 times ULN (≤ 5.0 times ULN if liver metastases are present)
* Bilirubin ≤ 1.5 times ULN (≤ 2.0 times ULN if liver metastases are present)
* Creatinine < 1.8 mg/dL
* Urine dipstick indicating 0-1+ protein

  * If dipstick reading is ≥ 2+, a 24-hour urine collection must demonstrate < 1 g of protein
* Prothrombin Time and International Normalized Ratio (PT/INR) ≤ 1.5 unless the patient is on therapeutic doses of warfarin, in which case the following criteria must be met:

  * Patient must have an in-range INR (between 2 and 3) on a stable dose of warfarin
  * Patient must not have active bleeding or a pathologic condition that is associated with a high risk of bleeding
* Patients with a history of non-colorectal malignancies must be disease free for ≥ 5 years prior to study entry and be deemed at low risk for recurrence
* Patients with the following cancers are eligible if diagnosed and treated within the past 5 years:

  * Carcinoma in situ of the colon
  * Melanoma in situ
  * Basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after the completion of study therapy
* No uncontrolled blood pressure (BP), defined as BP > 150/100 mm Hg
* No nonmalignant systemic disease that would preclude any of the study therapy drugs, compromise the safety of the patient, or inhibit the patient's ability to participate in the study, including any of the following:

  * New York Heart Association class III or IV cardiac disease
  * Myocardial infarction within the past 6 months
  * Unstable angina within the past 6 months
  * Symptomatic arrhythmia
* No transient ischemic attack or cerebrovascular accident within the past 6 months
* No symptomatic peripheral vascular ischemia within the past 6 months
* No arterial thrombotic event within the past 6 months
* No gastroduodenal ulcer(s) determined by endoscopy to be active
* No gastrointestinal perforation within the past 12 months
* No serious or nonhealing wound, skin ulcer, or bone fracture
* No significant traumatic injury within the past 28 days
* No significant episodes of acute bleeding requiring blood transfusion within the past 6 months
* No clinically significant (≥ grade 2) peripheral neuropathy (neurosensory or neuromotor toxicity)
* No pulmonary fibrosis or interstitial pneumonitis by chest x-ray
* No psychiatric or addictive disorders or other conditions that would preclude the patient from meeting study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy, radiation therapy, or surgery for this malignancy
* No prior endoscopic management of this malignancy other than biopsy, including endoscopic stent placement, fulguration, or laser treatment
* More than 30 days since prior investigational drugs
* More than 28 days since prior major surgical procedure or open biopsy
* More than 7 days since prior core biopsy or other minor procedure, excluding placement of a vascular access device
* No concurrent major surgery unrelated to intact primary colon cancer
* No concurrent radiotherapy
* No concurrent filgrastim (G-CSF) or pegfilgrastim as primary prophylaxis for neutropenia
* No concurrent halogenated antiviral agents
* No other concurrent investigational drugs
* No other concurrent antineoplastic agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (163):
- United States (163):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Scripps Cancer Center - San Diego, La Jolla, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care, Incorporated - Blue Ash, Cincinnati, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Started | 90
Completed | 86
Not Completed | 4
Not completed — Ineligible | 3
Not completed — No follow up data | 1

BASELINE CHARACTERISTICS:
Groups:
- Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Major Morbidity Related to the Intact Primary Tumor
Description: Cumulative incidence was used to compute percent probability of morbidity. Cumulative incidence at time t measures the probability of a participant having an event (i.e., Colonic bleeding, perforation, bowel obstruction, or fistula formation requiring surgery or resulting in patient death) over the given duration, t. It involves computing the probability of an event at any observed time (i.e., the number of new cases during a period divided by the number of subjects at risk) and multiplying these successive probabilities by any early computed probability to get the final estimate.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: probability of major morbidity (%)
Arm/Group | Arm 1: Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Number analyzed (Participants) | 86
probability of major morbidity (%) | 16.3 [7.6 to 25.1]

2. Secondary Outcome: Local Complications as Assessed by Colonic Obstruction Requiring Hospitalization (But Not Surgery) for Medical Management, Stent Placement, Laser Treatment, or Fulguration
Time Frame: Time from start of study through year 5
Reporting Status: Not Posted

3. Secondary Outcome: Local Complications as Assessed by Gastrointestinal Bleeding Requiring Transfusion But Not Requiring Surgery
Time Frame: Time from start of study through year 5
Reporting Status: Not Posted

4. Secondary Outcome: Local Complications as Assessed by Fistula Formation (Self-draining Enterocutaneous Fistula and Intra-abdominal Abscess Requiring Percutaneous Drainage) Not Requiring Surgery
Time Frame: Time from start of study through year 5
Reporting Status: Not Posted

5. Secondary Outcome: Local Complications as Assessed by Other Events Related to the Intact Primary Tumor Which Require Hospitalization But Not Surgery
Time Frame: Time from start of study through year 5
Reporting Status: Not Posted

6. Secondary Outcome: Serious Adverse Events (Grades 3, 4, and 5) as Defined by CTCAE v3.0
Time Frame: Time from start of study through year 5
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival as Measured by Death From Any Cause
Time Frame: Time from start of study through year 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an Adverse Event (AE) form.
Arm/Group | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/89
Other Adverse Events (participants affected / at risk) | 58/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab (N=89)
Diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin + Leucovorin + 5-Fluorouracil + Bevacizumab (N=89)
Abdominal pain (Gastrointestinal disorders) | 6
Anaphylaxis (Immune system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Fatigue (General disorders) | 14
Nausea (Gastrointestinal disorders) | 6
Neutrophil count decreased (Investigations) | 29
Peripheral sensory neuropathy (Nervous system disorders) | 14
Thromboembolic event (Vascular disorders) | 10
White blood cell decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less